CLINICAL TRIAL: NCT06700928
Title: The Effect of Different Attention-Focused Training on Physical Performance and Cognitive Function in Geriatric Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Müşerref Ebru ŞEN (Other)
Responsible Party: Sponsor-Investigator, Müşerref Ebru ŞEN, Principal Investigator, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/6463
Record Dates: First submitted 2024-11-14; First posted 2024-11-22 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-11

CONDITIONS: Geriatric Individuals; Cognitive Function; Physical Performance
Keywords: Geriatric individuals; Attention focus; Internal focus; External focus; Physical performance; Cognitive function

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Internal focus group (Experimental): After obtaining informed consent to participate in the study, all participants, regardless of group, will undergo an assessment by an experienced physiotherapist prior to group allocation. They will participate in exercise sessions lasting approximately 40 minutes, twice a week for 12 weeks in the internal focus group. A total of 24 sessions will be completed by each participant. Exercise sessions will be carried out by an experienced physiotherapist. Each training session will consist of warm-up (5 minutes), balance, transfer and reaching activities (10 minutes), internal focused walking (20 minutes) and cool-down (5 minutes) exercises.
  The first assessment will be made before the sessions start and the final assessment will be made after the 12-week exercise program.
  Interventions: Other: Internal focus training
- External focus group (Experimental): After obtaining informed consent to participate in the study, all participants, regardless of group, will undergo an assessment by an experienced physiotherapist prior to group allocation. They will participate in exercise sessions lasting approximately 40 minutes, twice a week for 12 weeks in the external focus group. A total of 24 sessions will be completed by each participant. Exercise sessions will be carried out by an experienced physiotherapist. Each training session will consist of warm-up (5 minutes), balance, transfer and reaching activities (10 minutes), external focused walking (20 minutes) and cool-down (5 minutes) exercises.
  The first assessment will be made before the sessions start and the final assessment will be made after the 12-week exercise program.
  Interventions: Other: External focus training
- No attention focus group (Experimental): After obtaining informed consent to participate in the study, all participants, regardless of group, will undergo an assessment by an experienced physiotherapist prior to group allocation. They will participate in exercise sessions lasting approximately 40 minutes, twice a week for 12 weeks in the no attention focus group. A total of 24 sessions will be completed by each participant. Exercise sessions will be carried out by an experienced physiotherapist. Each training session will consist of warm-up (5 minutes), balance, transfer and reaching activities (10 minutes), no attentional focus walking (20 minutes) and cool-down (5 minutes) exercises.
  The first assessment will be made before the sessions start and the final assessment will be made after the 12-week exercise program.
  Interventions: Other: No attentional focus training
- Control group (No Intervention): no-intervention

INTERVENTIONS:
Other: External focus training — External focus training
  Arms: External focus group
Other: Internal focus training — internal focus training
  Arms: Internal focus group
Other: No attentional focus training — no attentional focus training
  Arms: No attention focus group

SUMMARY:
The ability to walk safely and efficiently is crucial for older adults to maintain their independence and minimize the risk of falls. In healthy geriatric individuals, walking typically occurs as an automatic process involving motor skills, meaning the movement is generally performed with minimal conscious thought. However, attention can influence motor performance; a lack of focus or distraction can lead to loss of balance and increase the risk of falling during walking. The effects of attention focus on geriatric individuals remain uncertain. Therefore, this study aims to investigate the effects of different attention-focused training on physical performance and cognitive function in geriatric individuals. In this randomized controlled trial, 60 participants will be randomly assigned to four groups: the internal focus exercise group (n = 15), the external focus exercise group (n = 15), the no attention focus group (n = 15), and the control group (n = 15). The control group will consist of participants from a different institution to prevent contamination. Participants in the non-control groups will attend training sessions twice a week (approximately 40 minutes each) for 12 weeks. The experimental groups will complete a total of 24 exercise sessions. All training sessions will be conducted by an experienced physiotherapist. Pre- and post-assessments will be conducted. The sociodemographic characteristics of all participants will be assessed using a descriptive form. Participants' physical performance will be evaluated using the Short Physical Performance Battery (SPPB), the Stair Climbing Test, the Timed Up and Go Test (TUG), a static balance test (single-leg stance test), and a dynamic balance test (Berg Balance Scale). Cognitive function will be assessed using the Central Nervous System Vital Signs (CNSVS) Cognitive Performance and Attention Tests. Additionally, participants' walking will be analyzed using Kinect V2 camera-based software. The data collected from the study will be analyzed using SPSS (Statistical Program for the Social Sciences). Descriptive statistics will include frequencies, percentages, means, and standard deviations. For comparisons, the significance level (p) will be set at 0.05.

DETAILED DESCRIPTION:
Aging is an inevitable phase characterized by physiological and mental changes, including a decline in perception and awareness, as well as progressive deterioration of memory functions. According to the United Nations World Social Report (2023), the population aged 65 and older is expected to reach 1.6 billion by 2050.

With aging, motor performance, including balance, walking stability, postural stability, and movement speed, gradually declines. The literature indicates that one-third of individuals aged 65 and older experience a fall once or more per year, with the rate rising to 40% among those aged 85 and above. The risk of falling in older adults may be related to a decrease in the integration of physiological systems (cardiac, respiratory, and neuromuscular) that influence physical performance.

Physical performance is the objective measurement of an individual's ability to integrate various physiological systems (cardiac, respiratory, neuromuscular) to perform coordinated and effective movements. Due to its importance in evaluating mobility and overall physical well-being, it is considered a critical health indicator in older adults. The decline in physical performance can result from the complex interaction of physiological factors (e.g., declines in cardiovascular, musculoskeletal, and neuromuscular systems, leading to progressive loss of muscle mass and strength, reduced testosterone levels), clinical factors (e.g., depressive symptoms, multimorbidity, polypharmacy), lifestyle factors (e.g., physical activity levels), and sociodemographic factors (e.g., age, gender). This decline is evident not only in physical performance but also in cognitive function. With normal aging, the brain typically experiences shrinkage, a widely observed phenomenon, affecting both gray and white matter. This reduction in brain size is attributed to a decline in the development of dendrites, dendritic spines, axons, and synapses. As a result, cognitive abilities such as attention, memory, executive functions, language, and visuospatial skills decline with aging.

The decline in physical performance and cognitive function due to aging significantly impacts the ability to perform activities of daily living. The ability to walk safely and efficiently, which is essential for daily life, is necessary for older adults to maintain their independence and minimize the risk of falls. In healthy older adults, walking typically occurs with minimal conscious thought about the movement process. It is known that the focus of attention affects the performance of motor skills. The term "focus of attention" refers to the location of an individual's attention relative to the performance environment or task. This focus can be internal or external. An internal focus directs attention to the components of body movement during an action, whereas an external focus directs attention to the effect of the movement on the environment or the final goal. For example, during a ball throw, the individual may focus internally on the movement of the wrist, elbow, and shoulder, or externally on the ball and the target.

In recent years, various attention-focused approaches have been implemented to enhance functional and cognitive capacity in geriatric individualsProvidi. ng different attention-focus instructions to geriatric individuals has been shown to be an effective strategy for improving motor performance. A study examining the effects of internal focus, external focus, and no focus walking training during rehabilitation on conscious motor processing, balance, walking ability, and fear of falling in older adults at risk of falling found that focus reduced conscious motor processing while improving functional balance and walking (8). Furthermore, substantial evidence shows that using attention-focus methods results in improvements in physical performance. However, the effects of focus instructions on physical performance and cognitive function in geriatric individuals remain uncertain.

To address this gap in the literature, this study will investigate the effects of different attention-focus training on physical performance and cognitive function in geriatric individuals. We hypothesize that individuals who undergo attention-focused walking training during rehabilitation will demonstrate better physical performance and cognitive function compared to those who do not receive attention-focused walking training. Our study will provide data and contribute to filling this gap in the existing literature.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Willingness to participate in the study
* Ability to read and write
* Mini-Mental State Examination (MMSE) score > 24
* Ability to independently perform the tests administered as part of the study
* Ability to walk independently in the community (without a walking aid and able to walk at least 40 meters)

Exclusion Criteria:

* Presence of orthopedic, neurological, vestibular, cognitive, or other medical conditions that may affect the applicability of the assessment methods or training interventions used in the study
* History of myocardial infarction and/or coronary bypass surgery within the past year
* Severe visual or auditory impairments causing communication difficulties
* Polypharmacy (use of five or more medications per day)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The Short Physical Performance Battery (SPPB), stair climbing test, Timed Up and Go (TUG) test, Berg balance test, and single leg stance test | 12 weeks
  The Short Physical Performance Battery (SPPB), stair climbing test, Timed Up and Go (TUG) test, Berg balance test, and single leg stance test will be used to assess physical performance.
Central Nervous System Vital Signs (CNSVS) | 12 weeks
  The "Central Nervous System Vital Signs (CNSVS) Cognitive Performance and Attention Tests" will be administered to assess cognitive functions. CNSVS is an evaluation tool designed to examine the neurocognitive status of individuals aged 7 to 90. It consists of several subtests, including the Verbal Memory Test, Visual Memory Test, Finger Tapping Test, Symbol-Digit Coding Test, Stroop Test, Continuous Performance Test, and Attention Switching Test. In our study, scores obtained from these subtests will be utilized. To determine the extent of neurocognitive impairment, classification is made based on standard score points. According to this classification: >110 indicates high capacity, 90-110 indicates normal capacity, 80-89 indicates mild cognitive impairment, 70-79 indicates moderate cognitive impairment, and <70 indicates severe cognitive impairment.

SECONDARY OUTCOMES:
Gait analysis using Kinect V2 | 12 weeks
  The gait analysis of participants will be conducted using Kinect V2 camera-based software. This software is developed in the MATLAB environment and processes depth images to identify joint positions. It determines the corresponding joint position for each pixel in the depth image and calculates the accuracy of this position. This enables the detection and accuracy assessment of joint positions. Parameters such as gait symmetry, step length, step width, cadence, and speed will be evaluated.

IPD SHARING:
Plan to Share IPD: No
I think the data should be kept confidential.